CLINICAL TRIAL: NCT05639608
Title: EFFECT OF SCALING ON SERUM hsCRP LEVELS AND PERIODONTAL PARAMETERS IN SYSTEMICALLY HEALTHY WOMEN OF REPRODUCTIVE AGE GROUP WITH GINGIVITIS: AN INTERVENTIONAL STUDY
Brief Title: EFFECT OF SCALING ON SERUM hsCRP LEVELS AND PERIODONTAL PARAMETERS IN SYSTEMICALLY HEALTHY YOUNG WOMEN WITH GINGIVITIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: richa perio 2
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemically healthy females with gingivitis (Experimental): scaling will be done at baseline
  Interventions: Procedure: SCALING
- systemically and periodontally healthy females (No Intervention): data will be recorded at baseline and no intervention will be done

INTERVENTIONS:
Procedure: SCALING — SCALING WILL BE DONE AT BASELINE IN TEST GROUP.
  Arms: systemically healthy females with gingivitis

SUMMARY:
Gingivitis is a highly prevalent chronic bacterial disease in susceptible children, adults and the elderly, persisting for decades in subjects, and is an essential precursor of periodontitis. Several studies have shown periodontitis and subgingival P. gingivalis to be associated with increased C-reactive protein (CRP) levels and CRP has been implicated as a possible mediator of the association between periodontitis and several systemic diseases Limited data are available today addressing detrimental systemic effects of experimental or natural gingivitis as they have been rarely investigated. Results of various studies support the concept that gingivitis leads to systemic inflammation and that the level of systemic inflammatory markers increases proportionately with increase in gingival inflammation. It has also been seen that appropriate dental prophylaxis can also limit systemic markers of inflammation in subjects with natural gingivitis. Sex hormones have long been considered to play an influential role on periodontal tissues, bone turnover rate, wound healing and periodontal disease progression and can influence the cellular proliferation, differentiation and growth of keratinocytes and fibroblasts. Estrogen is mainly responsible for alterations in blood vessels and progesterone stimulates the production of inflammatory mediators. In addition, some micro-organisms found in the human mouth synthesize enzymes needed for steroid synthesis and catabolism. Sex hormones are neither necessary nor sufficient to produce gingival changes by themselves. However, they may alter periodontal tissue responses to microbial plaque and thus indirectly contribute to periodontal disease. (Markou). Till date, no study has been conducted assessing the serum hsCRP levels in females of reproductive age group with gingivitis. This study, thus, aims to assess the effect of scaling on serum hsCRP levels and periodontal parameters in systemically healthy women of reproductive age group with gingivitis.

DETAILED DESCRIPTION:
Gingivitis is a highly prevalent chronic bacterial disease in susceptible children, adults and the elderly, persisting for decades in subjects, and is an essential precursor of periodontitis. Several studies have shown periodontitis and subgingival P. gingivalis to be associated with increased C-reactive protein (CRP) levels and CRP has been implicated as a possible mediator of the association between periodontitis and several systemic diseases Limited data are available today addressing detrimental systemic effects of experimental or natural gingivitis as they have been rarely investigated. Results of various studies support the concept that gingivitis leads to systemic inflammation and that the level of systemic inflammatory markers increases proportionately with increase in gingival inflammation. It has also been seen that appropriate dental prophylaxis can also limit systemic markers of inflammation in subjects with natural gingivitis. Sex hormones have long been considered to play an influential role on periodontal tissues, bone turnover rate, wound healing and periodontal disease progression and can influence the cellular proliferation, differentiation and growth of keratinocytes and fibroblasts. Estrogen is mainly responsible for alterations in blood vessels and progesterone stimulates the production of inflammatory mediators. In addition, some micro-organisms found in the human mouth synthesize enzymes needed for steroid synthesis and catabolism. Sex hormones are neither necessary nor sufficient to produce gingival changes by themselves. However, they may alter periodontal tissue responses to microbial plaque and thus indirectly contribute to periodontal disease. (Markou). Till date, no study has been conducted assessing the serum hsCRP levels in females of reproductive age group with gingivitis. This study, thus, aims to assess the effect of scaling on serum hsCRP levels and periodontal parameters in systemically healthy women of reproductive age group with gingivitis.RESEARCH QUESTION What is the effect of scaling on serum hsCRP levels and periodontal parameters in systemically healthy women of reproductive age group with gingivitis?

* P -population-systemically healthy women,18-40 years of age having gingivitis.
* I-intervention- Scaling
* C -control/comparison- before and after scaling among systemically healthy women with gingivitis and also with systemically healthy women with healthy periodontium
* O -outcome- plaque index (PI), gingival index (GI), Bleeding on probing (BOP) and serum hsCRP levels
* T- time frame- 6 months

FINER

* F- feasibility- all the facilities required are present in the department.
* I-interesting-impact of scaling on systemic inflammation and periodontal status in women of reproductive age with gingivitis
* N-novelty- very little evidence available
* E-ethical-no ethical issues
* R-relevant-results of the study can help in further strengthening the link between local inflammatory burden and systemic inflammation by observing the effect of scaling on periodontium and systemic markers of inflammation and formulating recommendations for early periodontal care of the patients.

AIM - to assess the effect of scaling on serum hsCRP levels and periodontal parameters in systemically healthy women of reproductive age group with gingivitis.

OBJECTIVES - PRIMARY OBJECTIVES

1. Comparative evaluation of periodontal parameters [plaque index (PI),gingival index (GI), Bleeding on probing (BOP) ] and high sensitivity C reactive protein (hsCRP) levels in systemically healthy women having gingivitis before and after scaling.
2. Comparative evaluation of periodontal parameters [plaque index (PI),gingival index (GI), Bleeding on probing (BOP) ] and high sensitivity C reactive protein (hsCRP) levels among systemically healthy women having gingivitis and systemically healthy women with healthy periodontium.
3. To assess the association and correlation of periodontal parameters, anthropometric parameters and hsCRP levels in all patients.

SECONDARY OBJECTIVES

1. Comparative evaluation of Probing Depth (PD), Clinical attachment level (CAL)(in patients with reduced periodontium), anthropometric parameters of patients in both groups.
2. To compare and evaluate self-reported oral health quality of life questionnaire by the patients of both groups.

METHODOLOGY All the participants will be age and BMI matched. The present Randomized Controlled Trial will include 60 systemically healthy women in 2 groups.

Test group, n=30, systemically healthy women having gingivitis will receive oral hygiene instructions (OHI) and Scaling.

Control group, n=30, systemically healthy women having healthy periodontium will be assessed for hsCRP.

Periodontal and anthropometric parameters will be measured and sampling will be done at baseline, 3months and 6 months. Serum hsCRP levels will be assessed at baseline and also at 6 months in test group.

INTERVENTION- Scaling will be done with mechanical instruments and ultrasonic scalers at baseline. Oral hygiene instructions will be given verbally and brushing method will be demonstrated using a cast and a toothbrush.

ELIGIBILITY:
Inclusion Criteria:

* females of reproductive age group (18-40 yrs)
* BMI (18.5 - 24.9)
* presence of ≥20 natural teeth
* Healthy periodontium (for control group) defined as bleeding on probing at < 10% of sites, with pockets ≤3 mm, no probing attachment loss and no radiologic bone loss.
* Gingivitis (17) (for test group) Gingivitis (intact periodontium) is defined as bleeding on probing at ≥ 10% of sites, with pockets ≤3 mm, no probing attachment loss and no radiologic bone loss.

Gingivitis (reduced periodontium) is defined as bleeding on probing at ≥ 10% of sites with pockets ≤3 mm with possible probing attachment loss and possible radiologic bone loss.

Localized gingivitis is defined as 10-30% of bleeding sites. Generalized gingivitis is defined as more than 30% of bleeding sites.

Exclusion Criteria:

* history of androgen-secreting tumors, congenital adrenal hyperplasia and thyroid dysfunction
* nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, active cancer within the last past 5 years
* smokers and alcoholics
* history of systemic antibiotics or oral contraceptives usage within last 3 months
* periapical pathology or oral inflammatory conditions other than gingivitis.
* any periodontal treatment within 6 months prior to study Patients with pockets ≥ 3 mm and probing attachment loss shall be excluded, hence, radiographic examination will not be needed.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — females of reproductive age group shall be recruited
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
bleeding on probing | 6 months
  bleeding on probing will be measured on 6 sites per tooth in all the teeth
gingival index | 6 months
  gingival index will be measured on 4 sites per tooth in all the teeth
plaque index | 6 months
  plaque index will be measured on 4 sites per tooth in all the teeth
serum high sensitivity c reactive protein | 6 months
  serum high sensitivity C reactive protein will be measured at baseline and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richa Verma, BDS, Principal Investigator — Post Graduate Institute of Dental Sciences
Locations (2):
- India (2):
  - Post Graduate Institute of Dental Sciences, Rohtak, Haryana
  - Shikha Tewari, Rohtak, Haryana